CLINICAL TRIAL: NCT00512811
Title: Furosemide Inhalation in Dyspnea of Mustard Gas Exposed Patients: a Double-Blind Randomized Study
Brief Title: Furosemide Inhalation in Dyspnea of Mustard Gas Exposed Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 121a25
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Bronchiolitis
Keywords: furosemide; inhalation; dyspnea; spirometry; mustard gas; bronchiolitis; sulfur mustard
MeSH Terms: conditions — Bronchiolitis; Respiratory Aspiration; Dyspnea | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: furosemide

SUMMARY:
to assess the efficacy of inhaled furosemide in mustard gas exposed patients with acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of exposure to sulfur mustard with a complaint of dyspnea

Exclusion Criteria:

* A contraindication for furosemide use;
* An accompanying disease in which other drugs effective for dyspnea were used

Ages: 32 Years to 83 Years | Sex: Male
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
effect of furosemid inhalation on dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ghanei, MD, Study Chair — Research Center of Chemical Injuries, Baqiyatallah Medical Science University, Tehran, Iran
Locations (1):
- RCCI, Tehran, Tehran Province, Iran